CLINICAL TRIAL: NCT06048289
Title: Prospective Observational Study on Prediction of Response to First-line Immunotherapy in Patients With Biliary Tract Tumors
Brief Title: Prospective Observational Study to Predict the Response of Biliary Tract Tumors to Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Principal Investigator, Zhejiang Cancer Hospital
Other Study IDs: IRB-2020-404
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Biliary Tract Tumor; Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunotherapy combined with chemotherapy
  Interventions: Other: Blood samples, tumor biopsy specimens will be collected

INTERVENTIONS:
Other: Blood samples, tumor biopsy specimens will be collected — Blood samples, tumor biopsy specimens at baseline will be collected

SUMMARY:
A prospective, observational study to explore multidimensional biomarkers for predicting the efficacy of immunotherapy In biliary tract tumors

DETAILED DESCRIPTION:
Patient with unresectable advanced or metastatic biliary tract tumors will be enrolled and plan to receive PD-1/PD-L1 inhibitors combined with chemotherapy as first-line treatment. To explore the biomarkers, tumor tissues, acquired from puncture biopsies at baseline, will be collected and investigated by genomic panel sequencing , transcriptome sequencing, and mIHC. Meanwhile, baseline peripheral blood and feces were also collected for detection of plasma proteins, genomes, and metagenomes. Finally, the investigators will analysis and explore predictive biomarkers of immunotherapy in biliary tract tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old;
2. Imaging evaluation indicates unresectable advanced or metastatic biliary tract tumors (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder carcinoma);
3. Confirmed as adenocarcinoma by histology;
4. Has not received systemic therapy in the past (patients who have not progressed within six months after the completion of neoadjuvant therapy or adjuvant therapy can be enrolled);
5. At least one measurable lesion according to RECIST 1.1 standard;
6. Plan to receive PD-1/PD-L1 inhibitors combined with chemotherapy as first-line treatment;
7. Sign informed consent, has good compliance and can cooperate with follow-up.

Exclusion Criteria:

1. Suffering from other active malignant tumors within 5 years or simultaneously; Unable to collect baseline plasma or tissue samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a pathological diagnosis of biliary tract tumors who have agreed to receive first-line PD-1/PD-L1 inhibitors combined with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-14 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Identifying predictive biomarkers of immunotherapy response | 1 year
  ldentifying predictive biomarkers of immunotherapy response by detecting differences in genome and transcriptome sequencing between responder and non-responder patients

CONTACTS AND LOCATIONS:
Overall Officials: Biospecimen Retention Ying, Dr, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No